CLINICAL TRIAL: NCT00652379
Title: Co-treatment With Pegvisomant and a Somatostatin Analogue (SA) in SA-responsive Acromegalic Patients: Impact on Insulin Sensitivity, Glucose Tolerance, and Pharmacoeconomics
Brief Title: Co-treatment With Pegvisomant and a Somatostatin Analogue (SA) in SA-responsive Acromegalic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Aarhus University Hospital (Other); The Research Council for Health and Disease, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH-2007-228; 2007-005244-25 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-04-03 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Acromegaly; Insulin Resistance; Impaired Glucose Tolerance
Keywords: Acromegaly; Insulin sensitivity; Glucose tolerance; Body composition; Growth Hormone
MeSH Terms: conditions — Acromegaly; Insulin Resistance; Glucose Intolerance | interventions — pegvisomant; Somatostatin; lanreotide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Co-treatment with Pegvisomant (15-30 mg twice a week) and a 50 percent reduced somatostatin-analog dose
  Interventions: Drug: Pegvisomant; Drug: Somatostatin analog (lanreotide or octreotide)
- 2 (Active Comparator): Somatostatin analog, unaltered dosage
  Interventions: Drug: Somatostatin analog (lanreotide or octreotide)

INTERVENTIONS:
Drug: Pegvisomant — Pegvisomant s.c 15-30 mg 2 times a week
  Other Names: Somavert
  Arms: 1
Drug: Somatostatin analog (lanreotide or octreotide) — Study arm 2: usual dosage of a somatostatin analog Study arm 1: half dosage of somatostatin analog

SUMMARY:
The purpose of this study is to investigate if co-treatment of acromegalic patients, who beforehand are considered well-controlled on SA monotherapy, with pegvisomant and SA will improve insulin sensitivity and glucose tolerance, and if these effects of co-treatment can be obtained at a neutral cost as compared to SA mono therapy.

Second to investigate body composition, substrate metabolism, symptoms, intrahepatic and intramyocellular fat.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Diagnosed with acromegaly
* Safe anticonceptive for fertile women
* Well controlled on somatostatin analog (a serum IGF-I within normal range a nadir GH < 0.5 µg/l.)

Exclusion Criteria:

* Pregnancy
* Liver disease
* Diabetes mellitus type I
* Magnetic or electronic implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 0 and after 24 weeks

SECONDARY OUTCOMES:
Glucose tolerance | 0 and after 24 weeks
Symptoms, QoL questionaire | 0, 12 and 24 weeks
Intrahepatic and intramyocellular fat | 0 and 24 weeks
Substrate metabolism | 0 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, MD Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology, Aarhus University Hospital, Aarhus C, Aarhus, Denmark